CLINICAL TRIAL: NCT01451528
Title: The Efficacy and Safety of Allogeneic Umbilical Cord Blood Therapy for Chronic Traumatic Brain Injury Patients
Brief Title: Allogeneic Umbilical Cord Blood Therapy for Chronic TBI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The research fund, which is yet to be raised and expected to take for a while
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, MinYoung Kim, M.D., Associate Professor, Bundang CHA Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBIUCB; 2011-141 (Other: IRB of CHA Bundang Medical Center)
Record Dates: First submitted 2011-10-11; First posted 2011-10-13 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Traumatic Brain Injury
Keywords: Umbilical Cord Blood; Allogeneic; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Allogeneic Umbilical Cord Blood (Experimental): Allogeneic Umbilical Cord Blood Transplantation
  Interventions: Biological: Allogeneic Umbilical Cord Blood

INTERVENTIONS:
Biological: Allogeneic Umbilical Cord Blood — Allogeneic Umbilical Cord Blood Transplantation via Intravenous or Intraarterial route
  Other Names: Umbilical Cord Blood

SUMMARY:
This open label trial is conducted to investigate the efficacy and safety of umbilical cord blood therapy for chronic traumatic brain injury patients.

The study hypothesis is that the participants will show significant improvement in cognition and function after Umbilical cord blood (UCB) transplantation.

DETAILED DESCRIPTION:
Traumatic brain injury patients have been increasing due to various accidents. After acute therapeutic intervention, rehabilitation is the conventional main treatment with medication. However, in chronic stage, there seems to be some limitation in obtaining functional improvement in spite of comprehensive rehabilitation. Cell therapy like Umbilical cord blood (UCB) transplantation has showed promising results in many animal studies. The mechanism of such neurological improvement is not fully understood. Stem cells included in UCB are expected to secrete neurotrophic factors to enhance brain function. In addition, anti-inflammatory effects of UCB are suggested. Autologous UCB are not available in most of the cases in fact. The aim of this clinical trial is to determine the safety and efficacy of allogeneic UCB.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Traumatic Brain Injury Patient (onset duration: over 6 months)
* Glasgow Outcome Scale: 2, 3, 4, 5

Exclusion Criteria:

* High risk of pneumonia or renal function deterioration after immunosuppressant
* Possibility of drug hypersensitivity which is related to this study remedy
* Intractable seizure disorder
* Poor cooperation of guardian,including inactive attitude for rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Short-term Memory Function | Baseline - 6 months

SECONDARY OUTCOMES:
Changes in Global Outcome | Baseline - 6 months
Changes in Intelligence | Baseline - 6 months
Changes in Frontal Lobe Function | Baseline - 6 months
Changes in Traumatic Brain Injury-related Symptoms | Baseline - 6 months
Changes in Attention | Baseline - 6 months
Changes in Behavior | Baseline - 6 months
Changes in Emotion and Personality | Baseline - 6 months
Changes in Motor Function and Activities of Daily Living | Baseline - 6 months
Changes in Brain Structure | Baseline - 6 months
Changes in Brain Glucose Metabolism | Baseline - 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Minyoung Kim, M.D., Ph.D., Principal Investigator — CHA University
Locations (1):
- CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do, South Korea